CLINICAL TRIAL: NCT01045824
Title: The Genetic Study of Longitudinal Brain Function Among Schizophrenic Patients With Family History
Brief Title: Family-based Genetic Long-term Study of Brain Function in Schizophrenia
Acronym: FamilySchizo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: IRB TCVGH, Taichung Veterans General Hospital
Other Study IDs: C08202
Record Dates: First submitted 2010-01-06; First posted 2010-01-11 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Schizophrenia; Blooddraw; MRI
Keywords: Schizophrenia; DNA; MRI
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Family Based
Biospecimen Retention: Samples With DNA — 10-20cc of blood will be drawn for DNA analysis
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this research is to find out possible susceptible gene(s) in schizophrenic patients with family history and 5-year period functional changes of brain among the members of family, in order to further analysis factors and their interactions.

DETAILED DESCRIPTION:
Schizophrenia is a serious mental disease, highly family inheritable inclination. By means of traditional psychiatry diagnosis, genetics and long term brain change researches will help to unveil the secret of schizophrenia and other factors. The advantage of comparative gene hybridization is that chromosome copy number alterations can be detected; this technique has been widely applied in many researches, such as cancer, mental retardation screening and autism. As we known, we are the first one use this technique in chromosome abnormality research for family history schizophrenic patient, this study also is the first one to track the relationship of long term brain function alteration and chromosome abnormality in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1.Psychiatry doctor diagnosed who met the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for schizophrenia or schizoaffective disorder, family history, age older than 15 will be recruited for participation in this study. Participants agree and sign informed consent forms will eligible to participate this experiment.

2.10-20c.c blood will be drawn from the participants. 3.Participants need to understand procedures and assays of this experiment. 4.At least one psychiatry doctor interview needed, participants and their family voluntarily join this interview, approximately 30-45min.

Exclusion Criteria:

1. Participant can not understand procedures and assays of this experiment.
2. Participant has another major mental disease other than the inclusion criteria.
3. Participant has material abuse history, it could seriously influence diagnosis.
4. Participant has combination diseases, it could seriously influence diagnosis.
5. Psychopathy or psychosis can not be categorized in defined group.

Other considerations:

1. Participants, age fewer than 20 needs to their deputy guardians (parents) and their own consent altogether.
2. Participants who are inability needs to their deputy guardians (parents) and their own consent altogether.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Schizophrenia family
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2008-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tsuo-Hung Lan, MD., PhD., Study Director — Taichung Veterans General Hospital; Tsuo-Hung Lan, MD.,PhD, Study Director — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan, Taiwan